CLINICAL TRIAL: NCT02070302
Title: BOTOX® (Onabotulinumtoxin A) Injection(s) as a Treatment for Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benjamin Sucher (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Benjamin Sucher, Principal Investigator, Arizona Arthritis & Rheumatology Research, PLLC.
Organization: Arizona Arthritis & Rheumatology Research, PLLC. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 85700; 85700 (Other Grant/Funding Number: Allergan Sales. LLC)
Record Dates: First submitted 2014-02-20; First posted 2014-02-25 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin Type A (Active Comparator): After appropriate consent, each patient will receive 40 units of BOTOX® (onabotulinumtoxin A) divided into two injection sites of 20 units each into Opponens Pollicis (OP) and the Abductor Pollicis Brevis (APB)
  Interventions: Drug: Botulinum Toxin Type A
- Placebo (Placebo Comparator): .4cc/muscle of Normal saline will be injected into two injection sites each into Opponens Pollicis (OP) and the Abductor Pollicis Brevis (APB)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 40 units of BOTOX® (onabotulinumtoxin A) divided into two injection sites of 20 units each
  Other Names: Botox
  Arms: Botulinum Toxin Type A
Drug: Placebo — Placebo (Normal Saline) divided into 2 injections of .4cc each
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This study will be a prospective double blind controlled randomized trial of ten patients diagnosed with Carpal Tunnel Syndrome (CTS). The study will be completed at offices of medical practices in Arizona. Patients who meet inclusion criteria will be randomly distributed into two groups: a BOTOX® (onabotulinumtoxin A) injection group and a Normal Saline Injection (NS) (Placebo group). Each group will consist of five randomly assigned individuals.

DETAILED DESCRIPTION:
This is a pilot study, to assist with determining appropriate BOTOX® (onabotulinumtoxin A) dosing and injection locations in patients suffering from CTS.

Outcome measures will be obtained at follow-up at 6, 12, and 18 weeks post BOTOX® (onabotulinumtoxin A) injection and post saline injection using the same scales and instruments at baseline, namely Levine scale, JAMAR pinch dynamometer, EDX/NCS and NMUS. These measurements will be used to identify the effectiveness of BOTOX® (onabotulinumtoxin A) in decreasing thenar muscle strength, appropriate BOTOX® (onabotulinumtoxin A) injection dosing, and ability to decrease the inflammation, median nerve dysfunction, edema, symptoms of pain, numbness, and tingling often with associated with CTS.

ELIGIBILITY:
Inclusion Criteria:

* Patient history: evaluated using the Levine Scale for CTS, a self-administered questionnaire which assesses the function and severity of CTS.
* Physical Exam: including use of JAMAR pinch dynamometer to quantify initial baseline strength and confirm decreased pinch strength post injection to verify effective BOTOX® (onabotulinumtoxin A) injection.
* Electrodiagnostics (EDX): The following criteria would establish CTS through EDX namely baseline electromyogram (EMG) and nerve conduction studies (NCS): a) median nerve distal motor latency (DML) >4.3ms or >0.9ms above the ulnar nerve DML b) median distal sensory latency (DSL) to D-1 >2.9ms or >0.4ms above radial nerve D-1 DSL. c) median D-2 DSL >3.7ms or >0.4ms above ulnar nerve D-5 DSL (5). d) median mixed nerve palm-to-wrist latency (at 8cm) >2.2ms or >.3ms above ulnar mixed nerve palm-to-wrist latency (at 8cm).
* Imaging & Measurements (NMUS): Carpal tunnel images will be obtained in a transverse plane in both a neutral relaxed position at the level of the pisiform and longitudinally during neutral and Dynamic Stress Testing (DST) by a A Sonosite M-Turbo 6-13 MHz ultrasound system or another similar system (+ 2% accuracy). Measurements: Transverse images of the CT will measure the median nerve cross sectional area (CSA) at the level of the pisiform bone. CSA measurements greater than 11 mm2 are indicative of CTS. Borderline CSA measurements would require wrist forearm ratio (WFR) measurements to be a WFR > 1.5. Patients will need to have a CSA >11mm2, (or WFR >1.5) and show median nerve compression during DST of at least 30% to be included.

Exclusion Criteria:

* Patients with prior carpal tunnel surgery, prior history of BOTOX® (onabotulinumtoxin A) injection
* Steroid injection two months prior or three months after BOTOX® (onabotulinumtoxin A) CTS injection, median nerve denervation on needle EMG
* Major limb trauma or surgery, dysphagia
* Neuromuscular junction disorder (ie: Myasthenia gravis or Lambert-Eaton syndrome)
* Currently pregnant or breast feeding
* Patients with severe CTS identified by Levine scale >4, electrodiagnostics, and/or unable to meet the inclusion criteria as identified above would be excluded as participants in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Sucher, DO, Principal Investigator — Arizona Arthritis & Rheumatology Research
Locations (1):
- Arizona Arthritis & Rheumatology, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 10 patients with bilateral CTS, diagnosed by nerve conduction studies and NMUS (with crosssectional area measurements; and percentage of nerve compression measured during mechanical stress testing), divided into control and Onabot groups. Non-dominant hands were injected under ultrasound guidance with 40 units (0.4 cc) of Onabot or normal saline.
Groups:
- Botulinum Toxin Type A (Onabot): A prospective, randomized, double blind pilot study of patients with bilateral mild to moderate CTS, diagnosed by nerve conduction studies (NCS) and NMUS (with crosssectional area measurements; and percentage of nerve compression measured during mechanical stress testing). For 5 out of 10 subjects, non-dominant hands were injected under ultrasound guidance with 40 units of Onabot (0.4cc) divided equally into the abductor pollicis brevis and opponens pollicis muscles. Participants were evaluated with NMUS, NCS, Levine Scale (symptom severity and functional status), and Jamar dynamometer at baseline, 6, 12, and 18 weeks.
- Placebo: A prospective, randomized, double blind pilot study of 10 patients with bilateral mild to moderate CTS, diagnosed by nerve conduction studies (NCS) and NMUS (with crosssectional area measurements; and percentage of nerve compression measured during mechanical stress testing). Non-dominant hands were injected under ultrasound guidance with 40 units of 40 units of normal saline (0.4cc) divided equally into the abductor pollicis brevis and opponens pollicis muscles. Participants were evaluated with NMUS, NCS, Levine Scale (symptom severity and functional status), and Jamar dynamometer at baseline, 6, 12, and 18 weeks.
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A (Onabot) | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (17.9) | 52.3 (20.3) | 56.35 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Levine Symptom Severity Scale Status at Weeks 6, 12,18.
Description: Patients with Levine score < 4 were included in the study. The score for this assessment can range from 11-55.
Time Frame: Baseline-Week 18
Population: Levine symptom severity scale is a measure of mean of median value calculated for both Onabot and Placebo groups based on patient answered questions. It ranges from 1 (no symptoms) to 5 (severe symptoms). This scale indicate how severe the CTS symptoms feel to the patient. Mean values (std deviation) are reported both Onabot and Placebo groups.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 5 | 5
Scores on a scale
  Visit 2-Week 6 | 0.4 (6.8) | -3.2 (6.8)
  Visit 3-Week 12 | -4.2 (5.1) | -9.4 (8.3)
  Visit 4-Week 18 | -5.4 (8.7) | -6.8 (6.8)

2. Primary Outcome: Change From Baseline Levine Function Severity Scale Status at Weeks 6, 12,18.
Description: Patients with Levine score of < 4 were included in the study. The score for this assessment can range from 8-40
Time Frame: Baseline-Week 18
Population: Levine functional severity scale is a measure of mean of median value calculated for both Onabot and Placebo groups based on patient answered questions. This scale ranges from 1 (no symptoms) to 5 (severe symptoms). The function severity scale indicate interference of the symptoms on activities of daily living. Mean values reported for each group.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 5 | 5
Scores on a scale
  Visit 2-Week 6 | -1.0 (9.3) | -4.4 (11.9)
  Visit 3-Week 12 | -3.8 (4.8) | -9.6 (9.3)
  Visit 4-Week 18 | -4.0 (8.6) | -12.8 (6.1)

3. Primary Outcome: Change From Baseline in Median Nerve Compression on Neuromuscular Ultrasound at Week 6, Week 12, and Week 18.
Description: Neuromuscular ultrasound measures nerve compression (swelling) by cross sectional area of median nerve, in format % change from baseline.
Time Frame: Baseline to Week 18
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 5 | 5
% change
  Visit 2-Week 6 | -13.0 (15.3) | -20.2 (18.8)
  Visit 3-Week 12 | -15.9 (19.5) | -13.3 (9.4)
  Visit 4-Week 18 | -12.2 (17.8) | -4.7 (14.0)

4. Primary Outcome: Change From Baseline Electrodiagnostics Distal Sensory Median Nerve Latency at Week 6, Week 12, and Week 18.
Description: Latency is the interval between the stimulation of a muscle and the observed response, measuring conduction speed in milliseconds compared to baseline
Time Frame: Baseline, week 6, week 12, and week 18.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 5 | 5
milliseconds
  Visit 2-Week 6 | -0.1 (0.4) | -0.1 (0.1)
  Visit 3-Week 12 | -0.3 (0.3) | 0.0 (0.1)
  Visit 4-Week 18 | -0.3 (0.3) | -0.1 (0.3)

5. Primary Outcome: Change From Baseline Electrodiagnostics Motor Median Nerve Latency at Week 6, Week 12, and Week 18.
Description: Latency is the interval between the stimulation of a muscle and the observed response measuring nerve conduction speed in milliseconds.
Time Frame: Baseline to Week 18
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 5 | 5
milliseconds
  Visit 2-Week 6 | -0.2 (0.3) | -0.1 (0.1)
  Visit 3-Week 12 | -0.4 (0.5) | -0.1 (0.2)
  Visit 4-Week 18 | -0.6 (0.5) | -0.1 (0.3)

6. Primary Outcome: Change From Baseline Jamar Pinch (Unrelated Dominant Hand - Mean Value of All Repetitions/Positions) at Weeks 6, 12,18.
Description: Mean value of one finger and two finger opposition pinch between 1st and 5th and 1st with 4th and 5th phalanges.
Time Frame: Baseline-Week 18
Measure: Mean (Standard Deviation); unit: Pounds of Force (LBF)
Arm/Group | Botulinum Toxin Type A | Placebo
Number analyzed (Participants) | 5 | 5
Pounds of Force (LBF)
  Visit 2-Week 6 | 1.1 (1.2) | 0.5 (1.2)
  Visit 3-Week 12 | 1.4 (0.5) | -0.1 (1.7)
  Visit 4-Week 18 | 1.4 (0.5) | 0.4 (1.2)

ADVERSE EVENTS:
Time Frame: 18 weeks
Groups:
- Botulinum Toxin Type A: At 18 weeks, mean distal motor latency changes of -0.6 ms (P-value = 0.078) in the Onabot group were noted; and distal sensory latency changes of -0.3ms in the Onabot group; less slowing. Decreased mean cross-sectional area of -2.2 mm2 (P-value =0.040) in Onabot group were noted; less nerve edema. Decreased percent compression of the median nerve during stress testing was -12.6% in Onabot group. Three subjects injected with Onabot demonstrated decreases in median distal motor latencies that were nearly significant (p-value<.1, >.05), Two had decreases in median distal sensory latencies, and some had decreases in cross-sectional area on NMUS that were nearly significant. One Onabot subject did not show improvement or changes in median distal latencies but remained stable while the non-injected hand worsened with increasing median distal latencies.
Arm/Group | Botulinum Toxin Type A | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Botulinum Toxin Type A (N=5) | Placebo (N=5)
Left Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to the study
Neck Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to the study
Right Hand Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Related to the study.
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash on Left Groin Area. Not related to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No